CLINICAL TRIAL: NCT02520284
Title: A Combined Phase 2/3, Double-Blind, Randomized, Placebo-Controlled, Induction and Maintenance Study Evaluating the Safety and Efficacy of GS-5745 in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: Safety and Efficacy of Andecaliximab (GS-5745) in Adults With Moderately to Severely Active Ulcerative Colitis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-326-1100; 2014-005217-24 (EudraCT Number)
Record Dates: First submitted 2015-08-07; First posted 2015-08-11 (Estimated); Results first posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — andecaliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Andecaliximab Every 2 Weeks (Experimental): Participants will receive andecaliximab 150 mg administered via subcutaneous (SC) injection alternating with matching placebo weekly for a total of 4 doses of andecaliximab. Based on Week 8 assessment results, participants will either continue in Blinded Maintenance Treatment phase or will be offered Open-Label andecaliximab 150 mg administered via SC injection weekly for up to Week 51.
  Interventions: Biological: Andecaliximab; Biological: Placebo
- Andecaliximab Weekly (Experimental): Participants will receive andecaliximab 150 mg administered via SC injection once weekly for a total of 8 doses. Based on Week 8 assessment results, participants will either continue in Blinded Maintenance Treatment phase or will be offered Open-Label andecaliximab 150 mg administered via SC injection weekly for up to Week 51.
  Interventions: Biological: Andecaliximab
- Placebo (Placebo Comparator): Participants will receive placebo matched to andecaliximab administered via SC injection once weekly for a total of 8 doses. Based on Week 8 assessment results, participants will either continue in Blinded Maintenance Treatment phase or will be offered Open-Label andecaliximab 150 mg administered via SC injection weekly for up to Week 51.
  Interventions: Biological: Andecaliximab; Biological: Placebo

INTERVENTIONS:
Biological: Andecaliximab — Andecaliximab 150 mg administered via SC injection
  Other Names: GS-5745
Biological: Placebo — Placebo matched to andecaliximab administered via SC injection
  Arms: Andecaliximab Every 2 Weeks; Placebo

SUMMARY:
The primary objectives of this study are as follows: 1) To evaluate the efficacy of andecaliximab to induce endoscopy, rectal bleeding, and stool frequency (EBS) clinical remission at Week 8 (Cohort 1); 2) To evaluate the efficacy of andecaliximab to maintain EBS clinical remission at Week 52 (Cohort 2); and 3) To evaluate the safety and tolerability of andecaliximab. The study will consist of 3 parts: Induction Phase (Cohort 1), Maintenance Phase (Cohort 2), and an optional Extended Treatment Phase.

ELIGIBILITY:
Key Inclusion Criteria:

* Ulcerative Colitis (UC) confirmed on endoscopy
* Moderately to severely active UC (Mayo Score 6-12)
* May be receiving oral 5-aminosalicylate (ASA), oral corticosteroid, azathioprine, 6-mercaptopurine (MP), or methotrexate
* Treatment failure with at least one of the following agents received: corticosteroids, immunomodulators, tumor necrosis factor-alpha (TNFα) antagonists, vedolizumab

Key Exclusion Criteria:

* Diagnose of Crohn's disease or indeterminate colitis
* Pregnant or lactating females
* Any chronic medical condition (including, but not limited to cardiac or pulmonary disease, alcohol or drug abuse)
* Exhibit severe UC / clinically significant active infection
* History of malignancy in the last 5 years

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (87):
- United States (33):
  - Dothan, Alabama
  - Wheat Ridge, Colorado
  - Lauderdale Lakes, Florida
  - Miramar, Florida
  - Winter Park, Florida
  - Zephyrhills, Florida
  - Chicago, Illinois
  - Topeka, Kansas
  - Louisville, Kentucky
  - Monroe, Louisiana
  - Ann Arbor, Michigan
  - Plymouth, Minnesota
  - St Louis, Missouri
  - Egg Harbor, New Jersey
  - New York, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Mentor, Ohio
  - Rochester, Ohio
  - Germantown, Tennessee
  - Hermitage, Tennessee
  - Arlington, Texas
  - Baytown, Texas
  - Houston, Texas
  - Irving, Texas
  - San Antonio, Texas
  - Southlake, Texas
  - Charlottesville, Virginia
  - Chesapeake, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Wauwatosa, Wisconsin
- Australia (4):
  - Footscray
  - Herston
  - Malvern
  - Melbourne
- Belgium (3):
  - Ghent
  - Leuven
  - Mouscron
- Pleven, Bulgaria
- Canada (2):
  - Victoria, British Columbia
  - Vaughan, Ontario
- Hradec Králové, Czechia
- Nantes, France
- Hungary (3):
  - Békéscsaba
  - Budapest
  - Debrecen
- Dublin, Leinster, Ireland
- Italy (2):
  - Rozzano
  - San Giovanni Rotondo
- Daugavpils, Latvia
- Amsterdam, Netherlands
- New Zealand (3):
  - Christchurch, Canterbury
  - Auckland
  - Wellington
- Poland (10):
  - Bialystok
  - Krakow
  - Lublin
  - Piaseczno
  - Poznan
  - Sopot
  - Środa Wielkopolska
  - Tychy
  - Warsaw
  - Wroclaw
- Romania (2):
  - Bucharest
  - Timișoara
- Russia (4):
  - Moscow
  - Novosibirsk
  - Rostov-on-Don
  - Saint Petersburg
- Trenčín, Slovakia
- Claremont, Western Cape, South Africa
- South Korea (2):
  - Seoul
  - Suwon
- Switzerland (2):
  - Basel
  - Bern
- Taichung, Taiwan
- Ukraine (5):
  - Kharkiv
  - Kyiv
  - Lviv
  - Odesa
  - Vinnitsa
- United Kingdom (3):
  - Cambridge
  - Oxford
  - Prescot

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in South Africa, Europe, North America, and Asia Pacific. The first participant was screened on 15 September 2015. The last study visit occurred on 22 November 2016.
Pre-assignment Details: 241 participants were screened.
Groups:
- Andecaliximab Every 2 Weeks: Blinded Induction Phase: Participants received andecaliximab 150 mg administered via subcutaneous (SC) injection alternating with matching placebo weekly for a total of 4 doses of andecaliximab.
  Blinded Maintenance Phase: Participants who achieved endoscopy, rectal bleeding, and stool frequency (EBS) clinical remission and/or Mayo Clinical Score (MCS) response, based on Week 8 assessments, continued to receive andecaliximab 150 mg administered via SC injection alternating with matching placebo weekly for up to approximately 40 weeks.
  Open-Label Maintenance Phase: Participants who achieved neither EBS clinical remission nor MCS response, based on Week 8 assessments, were offered open-label andecaliximab 150 mg administered via SC injection once weekly for up to approximately 41 weeks.
- Andecaliximab Weekly: Blinded Induction Phase: Participants received andecaliximab 150 mg administered via SC injection once weekly for a total of 8 doses.
  Blinded Maintenance Phase: Participants who achieved EBS clinical remission and/or MCS response, based on Week 8 assessments, continued to receive andecaliximab 150 mg administered via SC injection once weekly for up to approximately 33 weeks.
  Open-Label Maintenance Phase: Participants who achieved neither EBS clinical remission nor MCS response, based on Week 8 assessments, were offered open-label andecaliximab 150 mg administered via SC injection once weekly for up to approximately 34 weeks.
- Placebo: Blinded Induction Phase: Participants received placebo matched to andecaliximab administered via SC injection once weekly for a total of 8 doses.
  Blinded Maintenance Phase: Participants who achieved EBS clinical remission and/or MCS response, based on Week 8 assessments, continued to receive placebo matched to andecaliximab administered via SC injection once weekly for up to approximately 39 weeks.
  Open-Label Maintenance Phase: Participants who achieved neither EBS clinical remission nor MCS response, based on Week 8 assessments, were offered open-label andecaliximab 150 mg administered via SC injection once weekly for up to approximately 38 weeks.
Period: Blinded Induction Phase: Up to Week 8
Arm/Group | Andecaliximab Every 2 Weeks | Andecaliximab Weekly | Placebo
Started | 54 | 56 | 55
Completed | 52 | 52 (1 Participant completed Blinded Induction Phase but did not continue further in study.) | 53 (1 Participant completed Blinded Induction Phase but did not continue further in study.)
Not Completed | 2 | 4 | 2
Not completed — Adverse Event | 1 | 3 | 0
Not completed — Withdrew Consent | 1 | 1 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 1
Period: Blinded Maintenance Phase: Up to Week 51
Arm/Group | Andecaliximab Every 2 Weeks | Andecaliximab Weekly | Placebo
Started | 20 (Participants achieving EBS remission and/or MCS response continued in Blinded Maintenance Phase.) | 16 (Participants achieving EBS remission and/or MCS response continued in Blinded Maintenance Phase.) | 18 (Participants achieving EBS remission and/or MCS response continued in Blinded Maintenance Phase.)
Completed | 0 | 0 | 0
Not Completed | 20 | 16 | 18
Not completed — Study Terminated by Sponsor | 17 | 11 | 15
Not completed — Disease Worsening | 2 | 2 | 3
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Disposition Error | 0 | 2 | 0
Period: Open-Label MaintenancePhase: Upto Week51
Arm/Group | Andecaliximab Every 2 Weeks | Andecaliximab Weekly | Placebo
Started | 32 (Participants achieving neither EBS remission nor MCS response entered Open-Label Maintenance Phase.) | 35 (Participants achieving neither EBS remission nor MCS response entered Open-Label Maintenance Phase.) | 34 (Participants achieving neither EBS remission nor MCS response entered Open-Label Maintenance Phase.)
Completed | 0 | 0 | 0
Not Completed | 32 | 35 | 34
Not completed — Study Terminated by Sponsor | 25 | 29 | 28
Not completed — Withdrew Consent | 3 | 4 | 2
Not completed — Adverse Event | 2 | 1 | 3
Not completed — Investigator's Discretion | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug in the Blinded Induction Phase.
Groups:
- Andecaliximab Every 2 Weeks: Blinded Induction Phase: Participants received andecaliximab 150 mg administered via SC injection alternating with matching placebo weekly for a total of 4 doses of andecaliximab.
  Blinded Maintenance Phase: Participants who achieved EBS clinical remission and/or MCS response, based on Week 8 assessments, continued to receive andecaliximab 150 mg administered via SC injection alternating with matching placebo weekly for up to approximately 40 weeks.
  Open-Label Maintenance Phase: Participants who achieved neither EBS clinical remission nor MCS response, based on Week 8 assessments, were offered open-label andecaliximab 150 mg administered via SC injection once weekly for up to approximately 41 weeks.
- Total: Total of all reporting groups
Arm/Group | Andecaliximab Every 2 Weeks | Andecaliximab Weekly | Placebo | Total
Number analyzed (Participants) | 54 | 56 | 55 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (14.1) | 43 (13.2) | 43 (12.8) | 43 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 24 | 61
  Male | 35 | 38 | 31 | 104
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 48 | 48 | 45 | 141
  Race: Black | 4 | 3 | 3 | 10
  Race: Asian | 2 | 4 | 4 | 10
  Race: Native Hawaiian or Pacific Islander | 0 | 0 | 1 | 1
  Race: Not Permitted | 0 | 0 | 1 | 1
  Race: Other | 0 | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 | 0 | 2 | 2
  Ethnicity: Not Hispanic or Latino | 54 | 56 | 51 | 161
  Ethnicity: Not Permitted | 0 | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 4 | 2 | 1 | 7
  Hungary | 1 | 2 | 2 | 5
  United States | 20 | 20 | 21 | 61
  Czechia | 1 | 0 | 1 | 2
  Ukraine | 3 | 3 | 3 | 9
  United Kingdom | 2 | 2 | 2 | 6
  Switzerland | 0 | 2 | 0 | 2
  Russia | 2 | 4 | 4 | 10
  New Zealand | 0 | 3 | 1 | 4
  Canada | 0 | 2 | 3 | 5
  South Korea | 2 | 3 | 2 | 7
  Latvia | 1 | 0 | 0 | 1
  Netherlands | 0 | 1 | 0 | 1
  Belgium | 1 | 3 | 2 | 6
  Ireland | 0 | 1 | 0 | 1
  Taiwan | 0 | 1 | 0 | 1
  Poland | 11 | 4 | 8 | 23
  Italy | 0 | 2 | 2 | 4
  South Africa | 1 | 1 | 0 | 2
  Slovakia | 1 | 0 | 0 | 1
  Australia | 3 | 0 | 2 | 5
  Bulgaria | 1 | 0 | 0 | 1
  France | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: For Cohort 1, Percentage of Participants With EBS Clinical Remission at Week 8
Description: EBS clinical remission was defined as an endoscopic subscore of 0 or 1 (endoscopic subscore range: 0 to 3, where 0 = normal or inactive disease and 3 = severe disease [spontaneous bleeding, ulceration]); rectal bleeding subscore of 0 (rectal bleeding subscore range: 0 to 3, where 0 = no blood seen and 3 = blood alone passes); and at least a 1-point decrease in stool frequency from baseline to achieve a subscore of 0 or 1 (stool frequency subscore range: 0 to 3, where 0 = normal number of stools and 3 = at least 5 stools more than normal).
Time Frame: Week 8
Population: Full Analysis Set included all randomized participants who received at least 1 dose of study drug in the Blinded Induction Phase (Cohort 1).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Andecaliximab Every 2 Weeks | Andecaliximab Weekly | Placebo
Number analyzed (Participants) | 54 | 56 | 55
percentage of participants | 7.4 [2.1 to 17.9] | 1.8 [0.0 to 9.6] | 7.3 [2.0 to 17.6]

2. Secondary Outcome: For Cohort 1, Percentage of Participants With MCS Remission at Week 8
Description: The MCS was composed of subscores from endoscopy (range: 0 to 3, where 0 = normal or inactive disease and 3 = severe disease [spontaneous bleeding, ulceration]), rectal bleeding (range: 0 to 3, where 0 = no blood seen and 3 = blood alone passes), stool frequency (range: 0 to 3, where 0 = normal number of stools and 3 = at least 5 stools more than normal), and physician's global assessment (PGA). The PGA acknowledged the participant's daily recollection of abdominal discomfort and general sense of wellbeing, and other observations, such as physical findings and the participant's performance status. The PGA score ranged from 0 to 3 with higher score indicating the severe disease. The MCS remission was defined as a MCS of ≤ 2 points and no individual subscore > 1 point. Total score for MCS ranged from 0 to 12 (sum of all subscores), with higher scores indicating disease worsening.
Time Frame: Week 8
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Andecaliximab Every 2 Weeks | Andecaliximab Weekly | Placebo
Number analyzed (Participants) | 54 | 56 | 55
percentage of participants | 7.4 [2.1 to 17.9] | 1.8 [0.0 to 9.6] | 7.3 [2.0 to 17.6]

3. Secondary Outcome: For Cohort 1, Percentage of Participants With MCS Response at Week 8
Description: The MCS was composed of subscores from endoscopy (range: 0 to 3, where 0 = normal or inactive disease and 3 = severe disease [spontaneous bleeding, ulceration]), rectal bleeding (range: 0 to 3, where 0 = no blood seen and 3 = blood alone passes), stool frequency (range: 0 to 3, where 0 = normal number of stools and 3 = at least 5 stools more than normal), and PGA. The PGA acknowledged the participant's daily recollection of abdominal discomfort and general sense of wellbeing, and other observations, such as physical findings and the participant's performance status. The PGA score ranged from 0 to 3 with higher score indicating the severe disease. Total score for MCS ranged from 0 to 12 (sum of all subscores), with higher scores indicating disease worsening. The MCS response was defined as a MCS reduction of ≥ 3 points and at least 30% from baseline, with an accompanying decrease in rectal bleeding subscore of ≥ 1 point or an absolute rectal bleeding subscore of 0 or 1.
Time Frame: Week 8
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Andecaliximab Every 2 Weeks | Andecaliximab Weekly | Placebo
Number analyzed (Participants) | 54 | 56 | 55
percentage of participants | 46.3 [32.6 to 60.4] | 30.4 [18.8 to 44.1] | 30.9 [19.1 to 44.8]

4. Secondary Outcome: For Cohort 1, Percentage of Participants With Endoscopic Remission at Week 8
Description: Endoscopic remission was defined as endoscopic subscore of 0. Endoscopic subscore range: 0 to 3, where 0 = normal or inactive disease and 3 = severe disease (spontaneous bleeding, ulceration).
Time Frame: Week 8
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Andecaliximab Every 2 Weeks | Andecaliximab Weekly | Placebo
Number analyzed (Participants) | 54 | 56 | 55
percentage of participants | 3.7 [0.5 to 12.7] | 0.0 [0.0 to 6.4] | 5.5 [1.1 to 15.1]

5. Secondary Outcome: For Cohort 1, Percentage of Participants With Endoscopic Response at Week 8
Description: Endoscopic response was defined as endoscopic subscore of 0 or 1. Endoscopic subscore range: 0 to 3, where 0 = normal or inactive disease and 3 = severe disease (spontaneous bleeding, ulceration).
Time Frame: Week 8
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Andecaliximab Every 2 Weeks | Andecaliximab Weekly | Placebo
Number analyzed (Participants) | 54 | 56 | 55
percentage of participants | 18.5 [9.3 to 31.4] | 7.1 [2.0 to 17.3] | 14.5 [6.5 to 26.7]

6. Secondary Outcome: For Cohort 1, Percentage of Participants With Mucosal Healing as Determined by the Geboes Histologic Scoring System at Week 8
Description: Mucosal healing was defined as elimination of ulcers/erosion, elimination of crypt destruction, elimination of intraepithelial neutrophils, elimination of lamina propria neutrophils, and reduction in lamina propria chronic inflammatory cells to at most a mild increase. When measured by the Geboes histologic scoring system, it was the selection of the following combined scores of ≤ 3 for Grade 0 (Structural Architectural Change), ≤ 1 for Grade 1 (Chronic Inflammatory Infiltrate), ≤ 3 for Grade 2A (Lamina Propria Eosinophils), and 0 for Grade 2B (Lamina Propria Neutrophils), Grade 3 (Neutrophils in Epithelium), Grade 4 (Crypt Destruction), and Grade 5 (Erosion or Ulceration). Total Geboes histologic score ranged from 0 to 22, with higher scores indicating greater disease severity.
Time Frame: Week 8
Population: Participants in the Full Analysis Set who did not meet the mucosal healing definition at baseline were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Andecaliximab Every 2 Weeks | Andecaliximab Weekly | Placebo
Number analyzed (Participants) | 50 | 51 | 50
percentage of participants | 18.0 [8.6 to 31.4] | 13.7 [5.7 to 26.3] | 22.0 [11.5 to 36.0]

7. Secondary Outcome: For Cohort 1, Percentage of Participants With MCS Remission (Alternative Definition) at Week 8
Description: The MCS remission (alternative definition) was defined as a rectal bleeding (range: 0 to 3, where 0 = no blood seen and 3 = blood alone passes), stool frequency (range: 0 to 3, where 0 = normal number of stools and 3 = at least 5 stools more than normal), and PGA subscore (range: 0 to 3 with higher score indicating the severe disease) of 0, and an endoscopic subscore (range: 0 to 3, where 0 = normal or inactive disease and 3 = severe disease [spontaneous bleeding, ulceration]) of 0 or 1 for an overall MCS of ≤ 1. Total score for MCS ranged from 0 to 12 (sum of all subscores), with higher scores indicating disease worsening.
Time Frame: Week 8
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Andecaliximab Every 2 Weeks | Andecaliximab Weekly | Placebo
Number analyzed (Participants) | 54 | 56 | 55
percentage of participants | 1.9 [0.0 to 9.9] | 0.0 [0.0 to 6.4] | 0.0 [0.0 to 6.5]

ADVERSE EVENTS:
Time Frame: Blinded Induction Phase: First dose of study drug to Week 8; Blinded Maintenance Phase: First dose of study drug up to approximately 39 weeks plus 30 days; Open-Label Maintenance Phase: First dose of open-label andecaliximab up to approximately 41 weeks plus 30 days
Description: Safety Analysis Set included all participants who received at least 1 dose of study drug in the Blinded Induction Phase. Safety data was summarized by the study periods (Blinded Induction Phase, Blinded Maintenance Phase, and Open-Label Maintenance Phase).
Groups:
- Blinded Induction Phase: Andecaliximab Every 2 Weeks: Adverse events reported in this group occurred during the Blinded Induction Phase. Participants received andecaliximab 150 mg administered via SC injection alternating with matching placebo weekly for a total of 4 doses of andecaliximab.
- Blinded Induction Phase: Andecaliximab Every Weeks: Adverse events reported in this group occurred during the Blinded Induction Phase. Participants received andecaliximab 150 mg administered via SC injection once weekly for a total of 8 doses.
- Blinded Induction Phase: Placebo: Adverse events reported in this group occurred during the Blinded Induction Phase. Participants received placebo matched to andecaliximab administered via SC injection once weekly for a total of 8 doses.
- Blinded Maintenance Phase: Andecaliximab Every 2 Weeks: Adverse events reported in this group occurred during the Blinded Maintenance Phase. Participants who achieved EBS clinical remission and/or MCS response, based on Week 8 assessments, continued to receive andecaliximab 150 mg administered via SC injection alternating with matching placebo weekly for up to approximately 40 weeks.
- Blinded Maintenance Phase: Andecaliximab Every Week: Adverse events reported in this group occurred during the Blinded Maintenance Phase. Participants who achieved EBS clinical remission and/or MCS response, based on Week 8 assessments, continued to receive andecaliximab 150 mg administered via SC injection once weekly for up to approximately 33 weeks.
- Blinded Maintenance Phase: Placebo: Adverse events reported in this group occurred during the Blinded Maintenance Phase. Participants who achieved EBS clinical remission and/or MCS response, based on Week 8 assessments, continued to receive placebo matched to andecaliximab administered via SC injection once weekly for up to approximately 39 weeks.
- Open-Label Maintenance Phase From Andecaliximab Every 2 Weeks: Adverse events reported in this group occurred during the Open-Label Maintenance Phase. Participants who achieved neither EBS clinical remission nor MCS response, based on Week 8 assessments, were offered open-label andecaliximab 150 mg administered via SC injection once weekly for up to approximately 41 weeks.
- Open-Label Maintenance Phase From Andecaliximab Every Week: Adverse events reported in this group occurred during the Open-Label Maintenance Phase. Participants who achieved neither EBS clinical remission nor MCS response, based on Week 8 assessments, were offered open-label andecaliximab 150 mg administered via SC injection once weekly for up to approximately 34 weeks.
- Open-Label Maintenance Phase From Placebo: Adverse events reported in this group occurred during the Open-Label Maintenance Phase. Participants who achieved neither EBS clinical remission nor MCS response, based on Week 8 assessments, were offered open-label andecaliximab 150 mg administered via SC injection once weekly for up to approximately 38 weeks.
Arm/Group | Blinded Induction Phase: Andecaliximab Every 2 Weeks | Blinded Induction Phase: Andecaliximab Every Weeks | Blinded Induction Phase: Placebo | Blinded Maintenance Phase: Andecaliximab Every 2 Weeks | Blinded Maintenance Phase: Andecaliximab Every Week | Blinded Maintenance Phase: Placebo | Open-Label Maintenance Phase From Andecaliximab Every 2 Weeks | Open-Label Maintenance Phase From Andecaliximab Every Week | Open-Label Maintenance Phase From Placebo
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/56 | 0/55 | 0/20 | 0/16 | 0/18 | 0/32 | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/54 | 2/56 | 1/55 | 1/20 | 2/16 | 1/18 | 1/32 | 3/35 | 2/34
Other Adverse Events (participants affected / at risk) | 24/54 | 31/56 | 26/55 | 12/20 | 12/16 | 13/18 | 9/32 | 6/35 | 12/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinded Induction Phase: Andecaliximab Every 2 Weeks (N=54) | Blinded Induction Phase: Andecaliximab Every Weeks (N=56) | Blinded Induction Phase: Placebo (N=55) | Blinded Maintenance Phase: Andecaliximab Every 2 Weeks (N=20) | Blinded Maintenance Phase: Andecaliximab Every Week (N=16) | Blinded Maintenance Phase: Placebo (N=18) | Open-Label Maintenance Phase From Andecaliximab Every 2 Weeks (N=32) | Open-Label Maintenance Phase From Andecaliximab Every Week (N=35) | Open-Label Maintenance Phase From Placebo (N=34)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Blinded Induction Phase: Andecaliximab Every 2 Weeks (N=54) | Blinded Induction Phase: Andecaliximab Every Weeks (N=56) | Blinded Induction Phase: Placebo (N=55) | Blinded Maintenance Phase: Andecaliximab Every 2 Weeks (N=20) | Blinded Maintenance Phase: Andecaliximab Every Week (N=16) | Blinded Maintenance Phase: Placebo (N=18) | Open-Label Maintenance Phase From Andecaliximab Every 2 Weeks (N=32) | Open-Label Maintenance Phase From Andecaliximab Every Week (N=35) | Open-Label Maintenance Phase From Placebo (N=34)
Anaemia (Blood and lymphatic system disorders) | 4 | 4 | 2 | 3 | 1 | 0 | 0 | 1 | 3
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 5 | 1 | 0 | 1 | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 2 | 3 | 1 | 2 | 1 | 4 | 1 | 1 | 3
Dyschezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 3 | 0 | 0 | 0 | 2 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 3 | 1 | 1 | 1 | 2 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Injection site bruising (General disorders) | 1 | 4 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Injection site hypersensitivity (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 4 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 2 | 2 | 0 | 2 | 2 | 1 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Injection related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 1 | 3 | 3 | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 1 | 2 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 4 | 1 | 0 | 2 | 1 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Menstrual disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to early termination of the study, Week 52 data were not available, and therefore prespecified Week 52 analyses could not be conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years